CLINICAL TRIAL: NCT05956574
Title: Healthy Living: Incorporating Lifestyle Interventions to Encourage a Reduction in Body Weight.
Brief Title: Lifestyle Intervention for Healthy Change
Acronym: LIVE WELL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Madison Kindred, Assistant Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020021-2
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Overweight and Obesity
Keywords: physical activity; dietary intervention
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Exercise; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrigenomix (Experimental): Participants in this group will be asked to complete an oral swab at baseline. This swab will indicate their dietary needs based on their genetic composition. These personalized dietary needs will be shared with the participant; the participant will be encouraged to follow their dietary plan for the duration of the study. Participants in this group will also gradually increase their physical activity up to 300 min/week at 6 months.
  Interventions: Behavioral: Nutrigenomix, personalized dietary plan; Behavioral: Physical Activity; Behavioral: Behavioral counseling
- Control (Active Comparator): Participants in this group will receive a standard care dietary plan. They will also be asked to gradually increase their activity up to 300 min/week by 6 months.
  Interventions: Behavioral: Physical Activity; Behavioral: Behavioral counseling; Behavioral: Standard Dietary plan

INTERVENTIONS:
Behavioral: Nutrigenomix, personalized dietary plan — Personalized dietary plan.
  Arms: Nutrigenomix
Behavioral: Physical Activity — Participate in an exercise program to work up to 300 min/week of moderate-intensity activity.
Behavioral: Behavioral counseling — Review behavioral counseling videos and participate in worksheets to assist with behavioral change.
Behavioral: Standard Dietary plan — Receive a standard dietary plan
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effectiveness of a physician led, multi-disciplinary approach to treating obesity that incorporates nutrition (mainly, using genetics to identify appropriate food intake), exercise, and motivational counseling. The investigators plan to recruit overweight/obese (BMI>25) males and females to participate. Participants will be randomized to receive a personalized diet plan, or a standard care diet plan; both groups will participate in the exercise intervention. For a 6-month duration, both groups will be asked to improve their diet according to their dietary plan and participate in moderate-to-vigorous physical activity (gradual increase up to 300 min/week). The investigators intend to evaluate standard outcomes of weight loss, and assess for any predictors of positive outcomes. Following the six-month intervention, participants will complete a 3-month no contact phase. This no contact phase will provide insight into the effects of the study on weight loss maintenance. Our team also plans to address acceptability by providing evaluations to study participants and conducting interviews with a small subset of participants to improve the intervention for the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* BMI > 25 kg/m2
* No cardiopulmonary disease
* stable on medications for 3 months
* weight stable (+/-5 pounds) for the past 3 months
* Not pregnant or trying to get pregnant
* Owns a smartphone
* Able to walk unassisted
* Not on supplemental oxygen

Exclusion Criteria:

* Under the age of 18 years
* 40 years and older
* Unable to participate in an exercise program
* Currently pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Total body weight | 6-months
  Use of scale to measure total body weight

CONTACTS AND LOCATIONS:
Overall Officials: Madison Kindred, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No